CLINICAL TRIAL: NCT00359203
Title: ISSUE3: International Study on Syncope of Uncertain Etiology 3 Pacemaker Therapy for Patients With Asystolic Neurally-mediated Syncope
Brief Title: ISSUE3: International Study on Syncope of Uncertain Etiology 3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ISS3
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2015-09

CONDITIONS: Syncope
Keywords: syncope; implantable loop recorder
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dual chamber pacemaker (Placebo Comparator): Dual chamber pacemaker programmed ODO (switched OFF)
  Interventions: Device: Dual chamber pacemeker
- Dual chamber pacemeker (Active Comparator): Medtronic dual chamber pacemaker programmed ON and with Rate Drope Response programmed ON
  Interventions: Device: Dual chamber pacemeker

INTERVENTIONS:
Device: Dual chamber pacemeker
  Other Names: Any model of Medtronic pacemakers with Rate Drop Respons algorhythm:; K700, K900, Enpulse, Advisa, Versa

SUMMARY:
ISSUE 3 is a multi-center, prospective, randomised controlled double-blind study aimed to assess the effectiveness of pacemaker therapy for prevention of asystolic neurally-mediated syncope.

DETAILED DESCRIPTION:
In asystolic neurally-mediated syncope (NMS) documented by Implantable Loop recorder (ILR), ISSUE-2, an observational trial, showed that pacemaker was effective in reducing the 1-year first syncope recurrence rate from 33% rate before implant (ILR phase 1) to 5% rate after implant (phase 2). Moreover, the control non-asystolic group still continued to have a 41% recurrence rate after the first recurrence of syncope, thus supporting the conclusion that the reduction with pacemaker was due to the beneficial effect of pacemaker itself and not to other factors. However a formal controlled trial is needed to confirm these findings.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or certain neurally-mediated syncope, based on the Guidelines recently published by the Task Force on Syncope of the European Society of Cardiology 2,3 (Appendix 1);
* More than 3 syncope episodes in the last 2 years;
* Clinical presentation of syncope of sufficient severity requiring treatment initiation in the physician's and patient's judgement.
* Age > 40 years.
* Negative carotid sinus massage.
* Patients accept to have an ILR implantation.

Exclusion criteria:

* Carotid sinus hypersensitivity
* Suspected or certain heart disease and high likelihood of cardiac syncope:
* Symptomatic orthostatic hypotension diagnosed by standing blood pressure measurement;
* Loss of consciousness different from syncope (e.g. epilepsy, psychiatric, metabolic, drop-attack, TIA, intoxication, cataplexy);
* Subclavian steal syndrome;
* Psychologically or physically (due to any other illness) or cognitively unfit for participation in the study according to the opinion of the investigator;
* Patient compliance doubtful;
* Patient geographically or otherwise inaccessible for follow-up;
* Patient unwilling or unable to give informed consent;
* Life expectancy <1 year.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Brignole, MD, Principal Investigator — Ospedali del Tigullio, Lavagna
Locations (1):
- Medtronic Italia S.p.A., Rome, Italy

REFERENCES:
- [Derived] Brignole M, Menozzi C, Moya A, Andresen D, Blanc JJ, Krahn AD, Wieling W, Beiras X, Deharo JC, Russo V, Tomaino M, Sutton R; International Study on Syncope of Uncertain Etiology 3 (ISSUE-3) Investigators. Pacemaker therapy in patients with neurally mediated syncope and documented asystole: Third International Study on Syncope of Uncertain Etiology (ISSUE-3): a randomized trial. Circulation. 2012 May 29;125(21):2566-71. doi: 10.1161/CIRCULATIONAHA.111.082313. Epub 2012 May 7. PMID 22565936
- See also: ISSUE3 main results publication PubMed — http://www.ncbi.nlm.nih.gov/pubmed/22565936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2007 to April 2011, 89 out of 511 patients (pts) implanted with implantable loop recorder (ILR) documented an asystolic syncope of >=3 sec or a non-syncopal asystole of >= 6 sec, inclusion criteria to be implanted with a dual chamber pacemaker (PM) and randomized to PM on or PM off. 77 pts out of 89 eligible pts were randomized.
Pre-assignment Details: 12 out of 89 eligible pts refused randomization
Groups:
- Dual Chamber Pacemaker OFF: Implant dual chamber pacemaker programmed ODO (switched OFF)
- Dual Chamber Pacemeker ON: Implant dual chamber pacemaker programmed ON and with Rate Drope Response algorhythm programmed ON
Period: Overall Study
Arm/Group | Dual Chamber Pacemaker OFF | Dual Chamber Pacemeker ON
Started | 39 | 38
Completed | 39 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dual Chamber Pacemaker OFF | Dual Chamber Pacemeker ON | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 17 | 39
  >=65 years | 17 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12) | 63 (14) | 63 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 16 | 20 | 36
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 16 | 36
  Spain | 8 | 8 | 16
  Netherlands | 1 | 0 | 1
  Austria | 1 | 0 | 1
  Germany | 3 | 4 | 7
  Canada | 1 | 2 | 3
  France | 2 | 3 | 5
  Switzerland | 1 | 0 | 1
  United Kingdom | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Syncope Recurrence Rate
Description: Intention to treat analysis of percentage of patients with syncope recurrence at 2 years follow-up after study arm assignement
Time Frame: 2 years
Population: 77 patients implanted with dual chamber pacemaker: 39 patients randomized to pacemaker OFF and 38 patients randomized to pacemaker ON
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dual Chamber Pacemaker OFF | Dual Chamber Pacemeker ON
Number analyzed (Participants) | 39 | 38
percentage of participants | 57 [40 to 74] | 25 [13 to 45]
Statistical Analysis 1: Comparison: Dual Chamber Pacemaker OFF vs Dual Chamber Pacemeker ON; The analysis was designed to have 80% power to detect a 1-year absolute reduction of 25% in the risk of recurrence of first syncope in the Pm ON arm applying a log-rank test with a 2-sided significance level of 0.05. This analysis was planned as a comparison of the cumulative risk of syncope between the 2 groups with the use of a log-rank test; Test type: Superiority or Other; p = 0.04, Log Rank; The risk of syncope recurrence was based on HR obtained by means of the univarate Cox model, with the use of the Breslow method for ties; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.19 to 0.96] — numerator=pacemaker ON denominator=pacemaker OFF
Statistical Analysis 2: Comparison: Dual Chamber Pacemaker OFF vs Dual Chamber Pacemeker ON; Test type: Non-Inferiority or Equivalence — The analysis was designed to have 80% power to detect a 1-year absolute reduction of 25% in the risk of recurrence of first syncope in the treatment arm applying a log-rank test with a 2-sided significance level of 0.05; p = 0.039, Log Rank — For the final analysis the threshold of statistical significance was set at 0.04; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.19 to 0.96] — Numerator=pacemaker ON denominator=pacemaker OFF

ADVERSE EVENTS:
Arm/Group | Dual Chamber Pacemaker OFF | Dual Chamber Pacemeker ON
Serious Adverse Events (participants affected / at risk) | 3/39 | 3/38
Other Adverse Events (participants affected / at risk) | 0/39 | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Chamber Pacemaker OFF (N=39) | Dual Chamber Pacemeker ON (N=38)
Right ventricle lead dislodgment (Surgical and medical procedures) | 2 (2) | 0 (0)
Right atrium lead dislodgment (Surgical and medical procedures) | 0 (0) | 2 (2)
Subclavian vein thrombosis (Surgical and medical procedures) | 1 (1) | 0 (0)
Dead (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Chamber Pacemaker OFF (N=39) | Dual Chamber Pacemeker ON (N=38)
Atrial arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No